CLINICAL TRIAL: NCT02513160
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, 6-Week Clinical Study to Assess the Efficacy and Safety of Beclomethasone Dipropionate Delivered Via Breath-Actuated Inhaler (BAI) at 320 or 640 mcg/Day in Adolescent and Adult Patients 12 Years of Age and Older With Persistent Asthma
Brief Title: Study to Assess the Efficacy and Safety of Beclomethasone Dipropionate in Adolescent and Adult Patients 12 Years of Age and Older With Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BDB-AS-30039; 2015-002510-80 (EudraCT Number)
Record Dates: First submitted 2015-07-28; First posted 2015-07-31 (Estimated); Results first posted 2017-09-11 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Persistent Asthma
MeSH Terms: interventions — Bays; Albuterol; Procaterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Beclomethasone dipropionate BAI 320 (Experimental): Beclomethasone Dipropionate Delivered via Breath-Actuated Inhaler (BAI) at 320 mcg/day (40 mcg/inhalation, 4 inhalations twice daily)
  Albuterol/salbutamol hydrofluoroalkane (HFA) metered-dose inhaler (MDI) (90 mcg ex-actuator) or equivalent was supplied by the sponsor for use as rescue medication during the run-in and double-blind study periods.
  Interventions: Drug: Beclomethasone dipropionate via 320 mcg BAI; Drug: albuterol/salbutamol
- Beclomethasone dipropionate BAI 640 (Experimental): Beclomethasone Dipropionate Delivered via Breath-Actuated Inhaler (BAI) at 640 mcg/day (80 mcg/inhalation, 4 inhalations twice daily)
  Albuterol/salbutamol hydrofluoroalkane (HFA) metered-dose inhaler (MDI) (90 mcg ex-actuator) or equivalent was supplied by the sponsor for use as rescue medication during the run-in and double-blind study periods.
  Interventions: Drug: Beclomethasone Dipropionate 640; Drug: albuterol/salbutamol
- Beclomethasone dipropionate MDI 320 (Active Comparator): Beclomethasone dipropionate Metered Dose Inhaler (MDI) 320 mcg/day (40 mcg/inhalation, 4 inhalations twice daily)
  Albuterol/salbutamol hydrofluoroalkane (HFA) metered-dose inhaler (MDI) (90 mcg ex-actuator) or equivalent was supplied by the sponsor for use as rescue medication during the run-in and double-blind study periods.
  Interventions: Drug: albuterol/salbutamol; Drug: Beclomethasone dipropionate via 320 mcg MDI
- Placebo (Placebo Comparator): Pooled breath-actuated inhaler (BAI) or metered-dose inhaler (MDI) placebo groups. Participants were instructed to take 4 inhalations twice daily for 6 weeks.
  Albuterol/salbutamol hydrofluoroalkane (HFA) metered-dose inhaler (MDI) (90 mcg ex-actuator) or equivalent was supplied by the sponsor for use as rescue medication during the run-in and double-blind study periods.
  Interventions: Drug: Placebo; Drug: albuterol/salbutamol

INTERVENTIONS:
Drug: Beclomethasone Dipropionate 640 — Beclomethasone Dipropionate 640 mcg BAI
  Arms: Beclomethasone dipropionate BAI 640
Drug: Placebo — Placebo, taken in the morning and evening each day, was provided in matching BAI and MDI devices.
  The placebo devices were identical to the devices used to deliver active drug.
  Arms: Placebo
Drug: Beclomethasone dipropionate via 320 mcg BAI — Beclomethasone dipropionate treatment administered via breath-actuated inhaler (BAI) (320 mcg/day).
  Arms: Beclomethasone dipropionate BAI 320
Drug: albuterol/salbutamol — Each patient's current rescue medication was replaced with study-supplied albuterol/salbutamol hydrofluoroalkane (HFA) metered-dose inhaler (MDI) (90 mcg ex-actuator) or equivalent during the run-in and double-blind study periods.
  Other Names: ProAir®
Drug: Beclomethasone dipropionate via 320 mcg MDI — Beclomethasone dipropionate treatment administered via metered-dose inhaler (MDI) (320 mcg/day).
  Other Names: QVAR® Inhalation Aerosol
  Arms: Beclomethasone dipropionate MDI 320

SUMMARY:
The primary objective of this study is to evaluate the efficacy of beclomethasone dipropionate administered via BAI at a dose strength of 40 or 80 mcg per oral inhalation (320 or 640 mcg/day, respectively) compared with placebo treatment in patients with persistent asthma as assessed by the standardized baseline-adjusted trough morning (pre-dose and pre-rescue bronchodilator) forced expiratory volume in 1 second (FEV1) area under the effect curve from time 0 to 6 weeks (AUEC[0-6wk]).

DETAILED DESCRIPTION:
Run-In Period (Days -14 to Day -1): Participants were provided with single-blind placebo breath-actuated inhaler (BAI) or metered-dose inhaler (MDI) device for twice-daily use after appropriate training and demonstration of the proper technique. Participants discontinued their current asthma therapy for the duration of the study.

Treatment Period (Day 0 to Week 6): Participants were randomly assigned to treatment and device type through a qualified randomization service provider (ie, IRT). The interactive response technology (IRT) system stratified patients based on treatment at the time of screening visit, either inhaled corticosteroid (ICS) or non-corticosteroid (NCS). During the study, blinded persons were blinded to treatment (active or placebo) assigned but not device (BAI or MDI) assignment.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a diagnosis of asthma as defined by the NIH. The asthma diagnosis
* has been present for a minimum of 3 months and has been stable (defined as no exacerbations and no changes in medication) for at least 30 days.
* The patient has been maintained on stable doses of :

  * non-corticosteroid therapy
  * inhaled corticosteroid therapy
* Written informed consent/assent is obtained. For adult patients (18 years of age and older, or as applicable per local regulations), the written informed consent form (ICF) must be signed and dated by the patient before conducting any study-related procedure. For minor patients (ages 12 to 17 years, or as applicable per local regulations), the written ICF must be signed and dated by the parent/legal guardian and the written informed assent form must be signed and dated by the patient before conducting any study-related procedure.
* The patient is a male or female 12 years of age or older as of the visit when informed consent/assent is signed (screening or prescreening visit, as applicable). (Note: Age requirements are as specified or allowed by local regulations.)
* The patient is able to perform acceptable and repeatable spirometry
* The patient is able to use an electronic diary after training.
* The patient is able to use devices properly
* If female, patient is currently not pregnant, not breast feeding, nor attempting to become pregnant (for 30 days before the screening visit (SV) and throughout the duration of the study and for 30 days after patient's last study visit) or, is of childbearing potential and not sexually active, has a negative urine pregnancy test, and is willing to commit to using a consistent and acceptable method of birth control
* If male, the patient is willing to commit to an acceptable method of birth control for the duration of the study, is surgically sterile or exclusively has same-sex partner(s).
* The patient does not have any concomitant conditions or treatments that could interfere with study conduct, influence the interpretation of study observations/results, or put the patient at increased risk during the study as judged by the investigator.
* The patient/parent/legal guardian is capable of understanding the requirements, risks, and benefits of study participation, and, as judged by the investigator, capable of giving informed consent/assent and being compliant with all study requirements (eg, dose schedules, visit schedules, procedures, and record keeping).
* The patient, as judged by the investigator, is able to discontinue all asthma medications at the SV.

  * other criteria apply, please contact the investigator for more information

Exclusion Criteria

* Life-threatening asthma, defined as a history of asthma episode(s) requiring intubation and/or associated with hypercapnea, respiratory arrest or hypoxic seizures, asthma-related syncopal episode(s), or hospitalizations within the past year.
* The patient received systemic corticosteroids within 30 days before the SV (for asthma exacerbation or for other indications).
* The patient has participated in any investigational drug study as a randomized patient within the 30 days (starting at the final visit of that study) preceding SV (or prescreening visit, as applicable), or plans to participate in another investigational drug study at any time during this study.
* The patient has previously participated in a beclomethasone dipropionate breath-actuated inhaler (device) (BAI) study as a randomized patient.
* The patient has a known hypersensitivity to any corticosteroid or any of the excipients in the study drug or rescue medication formulation.
* The patient has been treated with any known strong cytochrome inhibitors during the study.
* The patient has been treated with any of the prohibited medications during the prescribed (per protocol) withdrawal periods before the SV.
* The patient currently smokes or has a smoking history of 10 pack years or more (a pack year is defined as smoking 1 pack of cigarettes/day for 1 year). The patient may not have used tobacco products within the past year (eg, cigarettes, cigars, chewing tobacco, or pipe tobacco).
* The patient has a suspected bacterial or viral infection of the upper or lower respiratory tract, sinus, or middle ear that has not resolved at least 2 weeks before the SV.
* The patient has a history of alcohol or drug abuse within 2 years preceding SV.
* The patient has had an asthma exacerbation requiring oral corticosteroids within 1 month before the SV, or has had any hospitalization for asthma within 3 months before SV.
* The patient has initiated immunotherapy (administered by any route) less than 90 days before the SV or had a dose escalation of immunotherapy less than 30 days before the SV.
* The patient is unable to tolerate or unwilling to comply with the required washout periods and withholding of all applicable medications.
* The patient has untreated oral candidiasis at SV. Patients with clinical visual evidence of oral candidiasis and who agree to receive treatment and comply with appropriate medical monitoring may enter the study.
* The patient is either an employee or an immediate relative of an employee of the clinical investigational center.
* A member of the patient's household is participating in the study at the same time. (However, after the enrolled patient completes or discontinues participation in the study, another patient from the same household may be screened).
* The patient has a disease/condition that, in the medical judgment of the investigator, would put the safety of the patient at risk through participation or that could affect the efficacy or safety analysis if the disease/condition worsened during the study.

  * other criteria apply, please contact the investigator for more information

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 713 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (75):
- United States (75):
  - Teva Investigational Site 13415, Peoria, Arizona
  - Teva Investigational Site 13389, Downey, California
  - Teva Investigational Site 13421, Huntington Beach, California
  - Teva Investigational Site 13434, Huntington Beach, California
  - Teva Investigational Site 13427, Los Angeles, California
  - Teva Investigational Site 13386, Mission Viejo, California
  - Teva Investigational Site 13394, Orange, California
  - Teva Investigational Site 13417, Riverside, California
  - Teva Investigational Site 13445, Rolling Hills Estates, California
  - Teva Investigational Site 13420, San Diego, California
  - Teva Investigational Site 13443, San Diego, California
  - Teva Investigational Site 13438, San Jose, California
  - Teva Investigational Site 13397, Centennial, Colorado
  - Teva Investigational Site 13454, Denver, Colorado
  - Teva Investigational Site 13404, Aventura, Florida
  - Teva Investigational Site 13458, Hialeah, Florida
  - Teva Investigational Site 13416, Miami, Florida
  - Teva Investigational Site 13440, Miami, Florida
  - Teva Investigational Site 13455, Miami, Florida
  - Teva Investigational Site 13431, Ormond Beach, Florida
  - Teva Investigational Site 13437, Sarasota, Florida
  - Teva Investigational Site 13425, Tallahassee, Florida
  - Teva Investigational Site 13450, Normal, Illinois
  - Teva Investigational Site 13448, River Forest, Illinois
  - Teva Investigational Site 13408, Lenexa, Kansas
  - Teva Investigational Site 13410, Baltimore, Maryland
  - Teva Investigational Site 13422, Bethesda, Maryland
  - Teva Investigational Site 13435, Wheaton, Maryland
  - Teva Investigational Site 13411, North Dartmouth, Massachusetts
  - Teva Investigational Site 13398, Plymouth, Minnesota
  - Teva Investigational Site 13429, Plymouth, Minnesota
  - Teva Investigational Site 13433, Columbia, Missouri
  - Teva Investigational Site 13432, Rolla, Missouri
  - Teva Investigational Site 13414, St Louis, Missouri
  - Teva Investigational Site 13430, St Louis, Missouri
  - Teva Investigational Site 13384, Bellevue, Nebraska
  - Teva Investigational Site 13392, Brick, New Jersey
  - Teva Investigational Site 13426, Ocean City, New Jersey
  - Teva Investigational Site 13419, Skillman, New Jersey
  - Teva Investigational Site 13388, Rochester, New York
  - Teva Investigational Site 13441, Hickory, North Carolina
  - Teva Investigational Site 13403, Raleigh, North Carolina
  - Teva Investigational Site 13405, Wilmington, North Carolina
  - Teva Investigational Site 13395, Canton, Ohio
  - Teva Investigational Site 13396, Cincinnati, Ohio
  - Teva Investigational Site 13436, Sylvania, Ohio
  - Teva Investigational Site 13423, Toledo, Ohio
  - Teva Investigational Site 13387, Oklahoma City, Oklahoma
  - Teva Investigational Site 13453, Eugene, Oregon
  - Teva Investigational Site 13439, Lake Oswego, Oregon
  - Teva Investigational Site 13402, Medford, Oregon
  - Teva Investigational Site 13412, Portland, Oregon
  - Teva Investigational Site 13391, Pittsburgh, Pennsylvania
  - Teva Investigational Site 13449, East Providence, Rhode Island
  - Teva Investigational Site 13456, Warwick, Rhode Island
  - Teva Investigational Site 13413, North Charleston, South Carolina
  - Teva Investigational Site 13390, Knoxville, Tennessee
  - Teva Investigational Site 13442, Knoxville, Tennessee
  - Teva Investigational Site 13400, Austin, Texas
  - Teva Investigational Site 13452, Boerne, Texas
  - Teva Investigational Site 13407, Dallas, Texas
  - Teva Investigational Site 13424, Dallas, Texas
  - Teva Investigational Site 13409, El Paso, Texas
  - Teva Investigational Site 13451, Houston, Texas
  - Teva Investigational Site 13399, New Braunfels, Texas
  - Teva Investigational Site 13393, San Antonio, Texas
  - Teva Investigational Site 13444, San Antonio, Texas
  - Teva Investigational Site 13446, San Antonio, Texas
  - Teva Investigational Site 13457, San Antonio, Texas
  - Teva Investigational Site 13459, San Antonio, Texas
  - Teva Investigational Site 13383, Waco, Texas
  - Teva Investigational Site 13401, South Burlington, Vermont
  - Teva Investigational Site 13385, Richmond, Virginia
  - Teva Investigational Site 13447, Richmond, Virginia
  - Teva Investigational Site 13428, Greenfield, Wisconsin

REFERENCES:
- [Derived] Kerwin EM, Hickey L, Small CJ. Relationship between handheld and clinic-based spirometry measurements in asthma patients receiving beclomethasone. Respir Med. 2019 May;151:35-42. doi: 10.1016/j.rmed.2019.03.010. Epub 2019 Mar 20. PMID 31047115
- [Derived] Ostrom NK, Raphael G, Tillinghast J, Hickey L, Small CJ. Randomized trial to assess the efficacy and safety of beclomethasone dipropionate breath-actuated inhaler in patients with asthma. Allergy Asthma Proc. 2018 Mar 9;39(2):117-126. doi: 10.2500/aap.2018.39.4115. Epub 2018 Jan 9. PMID 29317015

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1089 patients with asthma were screened for enrollment into this study at 67 study centers in the US.
Pre-assignment Details: Of the screened patients, 376 patients were not enrolled; 312 were excluded on the basis of inclusion/exclusion criteria, 19 patients withdrew consent, 10 patients were lost to follow-up before the baseline visit, 1 patient reported an adverse event before entering run-in and the reason for screen failure was "Other" for 34 patients.
Groups:
- Placebo: Pooled breath-actuated inhaler (BAI) and metered-dose inhaler (MDI) placebo groups. Participants were instructed to take 4 inhalations twice daily for 6 weeks. Albuterol/salbutamol hydrofluoroalkane (HFA) metered-dose inhaler (MDI) (90 mcg ex-actuator) or equivalent was supplied by the sponsor for use as rescue medication during the run-in and double-blind study periods.
- BAI 320 mcg/Day: Beclomethasone dipropionate breath-actuated inhaler (BAI), 4 inhalations (40 mcg/inhalation), twice daily for a total daily dose of 320 mcg for 6 weeks. Albuterol/salbutamol hydrofluoroalkane (HFA) metered-dose inhaler (MDI) (90 mcg ex-actuator) or equivalent was supplied by the sponsor for use as rescue medication during the run-in and double-blind study periods.
- BAI 640 mcg/Day: Beclomethasone dipropionate breath-actuated inhaler (BAI), 4 inhalations (80 mcg/inhalation), twice daily for a total daily dose of 640 mcg for 6 weeks. Albuterol/salbutamol hydrofluoroalkane (HFA) metered-dose inhaler (MDI) (90 mcg ex-actuator) or equivalent was supplied by the sponsor for use as rescue medication during the run-in and double-blind study periods.
- MDI 320 mcg/Day: Beclomethasone dipropionate metered-dose inhaler (MDI), 4 inhalations (40 mcg/inhalation), twice daily for a total daily dose of 320 mcg for 6 weeks. Albuterol/salbutamol hydrofluoroalkane (HFA) metered-dose inhaler (MDI) (90 mcg ex-actuator) or equivalent was supplied by the sponsor for use as rescue medication during the run-in and double-blind study periods.
Period: Run-In Period (Days -14 to Day -1)
Arm/Group | Placebo | BAI 320 mcg/Day | BAI 640 mcg/Day | MDI 320 mcg/Day
Started | 713 (Enrolled) | 0 | 0 | 0
Completed | 425 | 0 | 0 | 0
Not Completed | 288 | 0 | 0 | 0
Not completed — Inclusion criteria not met | 33 | 0 | 0 | 0
Not completed — Failure to meet randomization criteria | 214 | 0 | 0 | 0
Not completed — Exclusion criteria met | 6 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 20 | 0 | 0 | 0
Not completed — Site reached randomization limit | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 10 | 0 | 0 | 0
Period: Treatment Period (Day 0 to Week 6)
Arm/Group | Placebo | BAI 320 mcg/Day | BAI 640 mcg/Day | MDI 320 mcg/Day
Started | 107 (Randomized) | 108 (Randomized) | 105 (Randomized) | 105 (Randomized)
Completed | 101 | 104 | 104 | 103
Not Completed | 6 | 4 | 1 | 2
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 1
Not completed — Noncompliance | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 1 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Did not meet exclusion criteria | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized; safety analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BAI 320 mcg/Day | BAI 640 mcg/Day | MDI 320 mcg/Day | Total
Number analyzed (Participants) | 107 | 108 | 105 | 105 | 425
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (13.33) | 41.8 (14.29) | 42.6 (14.19) | 43.1 (16.04) | 41.7 (14.52)
Age, Customized [Count of Participants; unit: Participants]
  12-17 years | 8 | 2 | 4 | 7 | 21
  18-64 years | 98 | 101 | 94 | 85 | 378
  >=65 years | 1 | 5 | 7 | 13 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 68 | 67 | 59 | 260
  Male | 41 | 40 | 38 | 46 | 165
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 87 | 92 | 83 | 84 | 346
  Black | 15 | 12 | 19 | 17 | 63
  Asian | 3 | 1 | 0 | 1 | 5
  American Indian or Alaskan Native | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0 | 0
  Other | 1 | 3 | 3 | 3 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 89 | 90 | 93 | 88 | 360
  Hispanic or Latino | 18 | 18 | 12 | 17 | 65
Weight [Mean (Standard Deviation); unit: kg] | 84.06 (25.337) | 89.93 (24.719) | 85.71 (25.590) | 88.56 (23.820) | 87.07 (24.987)
Height [Mean (Standard Deviation); unit: cm] | 167.34 (10.138) | 169.30 (9.457) | 167.82 (8.753) | 169.14 (8.770) | 168.40 (9.308)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.909 (8.4253) | 31.315 (8.1551) | 30.327 (8.3470) | 30.944 (8.1645) | 30.625 (8.2624)
Duration of Asthma [Count of Participants; unit: Participants]
  <3 months | 0 | 0 | 0 | 0 | 0
  3 months to <6 months | 0 | 0 | 0 | 0 | 0
  6 months to <1 year | 0 | 1 | 0 | 0 | 1
  1 year to <5 years | 5 | 8 | 6 | 5 | 24
  5 years to <10 years | 6 | 11 | 7 | 8 | 32
  10 years to <15 years | 12 | 7 | 8 | 12 | 39
  >=15 years | 84 | 81 | 84 | 80 | 329
Current Asthma Therapy [Count of Participants; unit: Participants]
  Inhaled corticosteroid | 66 | 66 | 65 | 65 | 262
  Non-corticosteroid | 41 | 42 | 40 | 40 | 163

OUTCOME MEASURES:

1. Primary Outcome: Standardized Baseline-Adjusted Trough Morning Forced Expiratory Volume in One Minute (FEV1) Area Under the Effect Curve From Time Zero to 6 Weeks (AUEC(0-6wk))
Description: The primary efficacy variable was the standardized baseline-adjusted trough morning (pre-dose and pre-rescue bronchodilator) FEV1 AUEC(0-6wk). Pulmonary function measurements such as FEV1 were obtained electronically by spirometry at the randomization visit, each treatment visit (Weeks 2, 4 and 6) and any unscheduled visit (such as the early termination visit). The highest FEV1 value from 3 acceptable and 2 repeatable maneuvers (maximum of 8 attempts) was used. The least-square (LS) means, difference of LS means and its 95% confidence interval (CI), and p-value represent the results obtained from the analysis of covariance with covariate adjustment for baseline, sex, age, current asthma therapy, and treatment.
Time Frame: Baseline (Day 0 of Treatment Period), weeks 2, 4, 6
Population: The modified intent-to-treat (mITT) analysis set included all patients in the ITT analysis set and included the available data for those patients until they discontinued study drug treatment at treatment visit week 6 or last available study visit.
Measure: Least Squares Mean (Standard Error); unit: milliliters
Arm/Group | Placebo | BAI 320 mcg/Day | BAI 640 mcg/Day | MDI 320 mcg/Day
Number analyzed (Participants) | 105 | 105 | 104 | 103
milliliters | 62 (23.0) | 205 (23.2) | 212 (23.3) | 210 (23.0)
Statistical Analysis 1: Comparison: Placebo vs BAI 640 mcg/Day; A fixed-sequence multiple testing procedure was implemented to interpret the results from the primary analysis while controlling the family-wise error rate at 5%. The 640-mcg/day BAI dose was tested first. If the comparison to placebo resulted in p≤0.05, the 320-mcg/day BAI dose was then tested; Test type: Superiority or Other; p < 0.0001, ANCOVA — a priori threshold for significance of 0.05; Difference of LS means, 95% CI, and p-value represent ANCOVA results adjusted for baseline, sex, age, current asthma therapy, and treatment; LSM difference = 150, 95% CI 2-sided [86.8 to 213.2] — Active - placebo
Statistical Analysis 2: Comparison: Placebo vs BAI 320 mcg/Day; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — a priori threshold for significance of 0.05; [statistical method as in outcome 1, analysis 1]; LSM difference = 144, 95% CI 2-sided [80.7 to 206.6] — Active - placebo
Statistical Analysis 3: Comparison: Placebo vs MDI 320 mcg/Day; Test type: Superiority or Other; p < 0.0001, ANCOVA — a priori threshold for significance of 0.05. The p-value was not adjusted; Difference of LS means and 95% CI represent ANCOVA results adjusted for baseline, sex, age, current asthma therapy, and treatment; LSM difference = 148, 95% CI 2-sided [84.7 to 211.4] — Active - placebo

2. Secondary Outcome: Change From Baseline in Weekly Average of Daily Trough Morning Peak Expiratory Flow (PEF) Rate Over the 6-Week Treatment Period
Description: Change from baseline in the weekly average of daily trough morning (pre-dose and pre-rescue bronchodilator) PEF by handheld spirometer over the 6-week treatment period. PEF were determined twice daily, in the morning and in the evening, before administration of study drug or rescue medications. A handheld spirometer was provided to patients and used to determine the morning and evening PEF throughout the study. The spirometer was programmed to record the highest PEF obtained from 3 valid attempts. Baseline was defined as the average of recorded trough morning PEF assessments over the 7 days prior to the first dose of double-blind study treatment, including the morning assessment at the randomization visit. The LS means, difference of LS means and its 95% confidence interval, and p value are obtained from the mixed model for repeated measures analysis with covariate adjustment for baseline, sex, age, current asthma therapy, treatment, week, and treatment by week interaction.
Time Frame: Timeframes: Baseline (Day -7 to Day 0 which is part of the Run-in Period); Treatment Period from Day 0 up to 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters/minute
Arm/Group | Placebo | BAI 320 mcg/Day | BAI 640 mcg/Day | MDI 320 mcg/Day
Number analyzed (Participants) | 106 | 108 | 105 | 104
liters/minute | -10.0 (4.31) | 20.1 (4.30) | 11.9 (4.28) | 10.9 (4.28)
Statistical Analysis 1: Comparison: Placebo vs BAI 640 mcg/Day; Treatment comparisons began with am PEF for BAI 640 mcg/day vs placebo. If the p-value was ≤0.05, the next comparisons of interest were made 1) the next secondary outcome comparison for BAI 640 mcg/day vs placebo 2) the am PEF for BAI 320 mcg/day vs placebo. This procedure allowed for control of the Type I error for comparisons at a particular BAI treatment over the 5 secondary endpoints, as well as comparisons within an endpoint. It did not control the overall Type I error; Test type: Superiority or Other; p = 0.0003, mixed model for repeated measures — a priori threshold for significance of 0.05; MMRM analysis with covariates for baseline, sex, age, current asthma therapy, treatment, week, and treatment by week interaction; LSM difference = 21.9, 95% CI 2-sided [10.11 to 33.71] — Active - placebo
Statistical Analysis 2: Comparison: Placebo vs BAI 320 mcg/Day; Sequential order of analyses described in previous analysis; Test type: Superiority or Other; p < 0.0001, mixed model for repeated measures — a priori threshold for significance of 0.05; [statistical method as in outcome 2, analysis 1]; LSM difference = 30.1, 95% CI 2-sided [18.33 to 41.90] — Active - placebo
Statistical Analysis 3: Comparison: Placebo vs MDI 320 mcg/Day; Comparisons for MDI dose versus placebo for the secondary efficacy endpoints were used for assay sensitivity; Test type: Superiority or Other; p = 0.0006, mixed model for repeated measures — a priori threshold for significance of 0.05; [statistical method as in outcome 2, analysis 1]; LSM difference = 21.0, 95% CI 2-sided [9.14 to 32.83] — Active - placebo

3. Secondary Outcome: Change From Baseline in Weekly Average of Daily Trough Morning Forced Expiratory Volume in One Minute (FEV1) Rate Over the 6-Week Treatment Period
Description: Change from baseline in the weekly average of daily trough morning (pre-dose and pre-rescue bronchodilator) FEV1 by handheld spirometer over the 6-week treatment period. FEV1 were determined twice daily, in the morning and in the evening, before administration of study drug or rescue medications. A handheld spirometer was provided to patients and used to determine the morning and evening FEV1 throughout the study. The spirometer was programmed to record the highest FEV1 obtained from 3 valid attempts. Baseline was defined as the average of recorded trough morning FEV1 assessments over the 7 days prior to the first dose of double-blind study treatment, including the morning assessment at the randomization visit. The LS means, difference of LS means and its 95% confidence interval, and p value are obtained from the mixed model for repeated measures analysis with covariate adjustment for baseline, sex, age, current asthma therapy, treatment, week, and treatment by week interaction.
Time Frame: Baseline (Day -7 to Day 0 which is part of the Run-in Period); Treatment Period from Day 0 up to 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milliliters
Arm/Group | Placebo | BAI 320 mcg/Day | BAI 640 mcg/Day | MDI 320 mcg/Day
Number analyzed (Participants) | 106 | 108 | 105 | 104
milliliters | -8 (26.0) | 162 (25.8) | 135 (25.9) | 125 (25.8)
Statistical Analysis 1: Comparison: Placebo vs BAI 640 mcg/Day; Sequential order of analyses described in Outcome #2, analysis #1; Test type: Superiority or Other; p < 0.0001, mixed model for repeated measures — a priori threshold for significance of 0.05; [statistical method as in outcome 2, analysis 1]; LSM difference = 143, 95% CI 2-sided [71.7 to 214.1] — Active - placebo
Statistical Analysis 2: Comparison: Placebo vs BAI 320 mcg/Day; Sequential order of analyses described in Outcome #2, analysis #1; Test type: Superiority or Other; p < 0.0001, mixed model for repeated measures — a priori threshold for significance of 0.05; [statistical method as in outcome 2, analysis 1]; LSM difference = 170, 95% CI 2-sided [98.5 to 240.5] — Active - placebo
Statistical Analysis 3: Comparison: Placebo vs MDI 320 mcg/Day; Comparisons for MDI dose versus placebo for the secondary efficacy endpoints were used for assay sensitivity; Test type: Superiority or Other; p = 0.0003, mixed model for repeated measures — a priori threshold for significance of 0.05; [statistical method as in outcome 2, analysis 1]; LSM difference = 133, 95% CI 2-sided [61.3 to 204.3] — Active - placebo

4. Secondary Outcome: Change From Baseline in Weekly Average of Total Daily (24-Hour) Rescue Medication Use Over the 6-Week Treatment Period
Description: Change from baseline in the weekly average of total daily (24-hour) use of albuterol/salbutamol inhalation aerosol over weeks 1 through 6. Patients recorded the number of inhalations (puffs used) of rescue medication (albuterol/salbutamol HFA MDI [90 mcg ex-actuator] or equivalent) each morning and evening in the diary. The average number of daily inhalations over the 7 days before the randomization visit was the baseline value and was compared with the rescue medication use during the 6-week treatment period.
Time Frame: Baseline (Day -7 to Day 0 which is part of the Run-in Period); Treatment Period from Day 0 up to 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: number of inhalations
Arm/Group | Placebo | BAI 320 mcg/Day | BAI 640 mcg/Day | MDI 320 mcg/Day
Number analyzed (Participants) | 106 | 108 | 105 | 104
number of inhalations | 0.37 (0.140) | -0.73 (0.139) | -0.66 (0.140) | -0.66 (0.139)
Statistical Analysis 1: Comparison: Placebo vs BAI 640 mcg/Day; Sequential order of analyses described in Outcome #2, analysis #1; Test type: Superiority or Other; p < 0.0001, mixed model for repeated measures — a priori threshold for significance of 0.05; [statistical method as in outcome 2, analysis 1]; LSM difference = -1.02, 95% CI 2-sided [-1.408 to -0.640] — Active - placebo
Statistical Analysis 2: Comparison: Placebo vs BAI 320 mcg/Day; Sequential order of analyses described in Outcome #2, analysis #1; Test type: Superiority or Other; p < 0.0001, mixed model for repeated measures — a priori threshold for significance of 0.05; [statistical method as in outcome 2, analysis 1]; LSM difference = -1.10, 95% CI 2-sided [-1.482 to -0.717] — Active - placebo
Statistical Analysis 3: Comparison: Placebo vs MDI 320 mcg/Day; Comparisons for MDI dose versus placebo for the secondary efficacy endpoints were used for assay sensitivity; Test type: Superiority or Other; p < 0.0001, mixed model for repeated measures — a priori threshold for significance of 0.05; [statistical method as in outcome 2, analysis 1]; LSM difference = -1.03, 95% CI 2-sided [-1.415 to -0.643] — Active - placebo

5. Secondary Outcome: Change From Baseline in Weekly Average of Total Daily Asthma Symptom Score Over the 6-Week Treatment Period
Description: Asthma symptom scores were recorded in the patient's diary each morning and evening before determining FEV1 and PEF and before administration of study or rescue medications. The Daytime Symptom Score was recorded in the evening on a scale of 0 (No symptoms during the day) to 5 (Symptoms so severe that I could not go to work or perform normal daily activities) plus the Nighttime Symptom Score in the morning on a scale of 0 (No symptoms during the night) to 4 (Symptoms so severe that I did not sleep at all) for a total score range of 0-9. Baseline was defined as the average of recorded daily asthma symptom scores (average of daytime and nighttime score) over the 7 days prior to the first dose of double-blind study treatment, including the morning assessment at the randomization visit. The LS means, difference of LS means and its 95% CI, and p value are obtained from the mixed model for repeated measures analysis with covariate adjustment for baseline, sex, age, current asth
Time Frame: Baseline (Day -7 to Day 0 which is part of the Run-in Period); Treatment Period from Day 0 up to 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | BAI 320 mcg/Day | BAI 640 mcg/Day | MDI 320 mcg/Day
Number analyzed (Participants) | 106 | 107 | 105 | 104
units on a scale | 0.06 (0.043) | -0.18 (0.043) | -0.26 (0.043) | -0.24 (0.043)
Statistical Analysis 1: Comparison: Placebo vs BAI 640 mcg/Day; Sequential order of analyses described in Outcome #2, analysis #1; Test type: Superiority or Other; p < 0.0001, mixed model for repeated measures — a priori threshold for significance of 0.05; [statistical method as in outcome 2, analysis 1]; LSM difference = -0.32, 95% CI 2-sided [-0.440 to -0.203] — Active - placebo
Statistical Analysis 2: Comparison: Placebo vs BAI 320 mcg/Day; Sequential order of analyses described in Outcome #2, analysis #1; Test type: Superiority or Other; p < 0.0001, mixed model for repeated measures — a priori threshold for significance of 0.05; [statistical method as in outcome 2, analysis 1]; LSM difference = -0.25, 95% CI 2-sided [-0.365 to -0.128] — Active - placebo
Statistical Analysis 3: Comparison: Placebo vs MDI 320 mcg/Day; Comparisons for MDI dose versus placebo for the secondary efficacy endpoints were used for assay sensitivity; Test type: Superiority or Other; p < 0.0001, mixed model for repeated measures — a priori threshold for significance of 0.05; [statistical method as in outcome 2, analysis 1]; LSM difference = -0.30, 95% CI 2-sided [-0.423 to -0.185] — Active - placebo

6. Secondary Outcome: Count of Participants Withdrawn From Study Drug Treatment Due to Meeting Stopping Criteria for Worsening Asthma
Description: Number of participants who were withdrawn from study drug due to worsening asthma. Alert criteria for individual patients with worsening asthma were designed to ensure patient safety. The investigator determined whether the patient's overall clinical picture was consistent with worsening asthma and if the patient should be withdrawn from study drug treatment (but not the study) and be placed on appropriate asthma therapy in the interest of patient safety. An example of an alert criteria is:
  * Morning FEV1 by handheld spirometer as measured at home falls below the FEV1 stability limit (FEV1 <80%) as calculated at the screening visit for the Run-in Period and at the randomization visit (Day 0) for the Treatment Period on 4 or more days out of any 7-day period.
Time Frame: Day 0 to Week 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BAI 320 mcg/Day | BAI 640 mcg/Day | MDI 320 mcg/Day
Number analyzed (Participants) | 107 | 108 | 105 | 105
Participants | 10 | 1 | 0 | 1
Statistical Analysis 1: Comparison: Placebo vs BAI 320 mcg/Day; Test type: Superiority or Other; p = 0.0058, Log Rank
Statistical Analysis 2: Comparison: Placebo vs BAI 640 mcg/Day; Test type: Superiority or Other; p = 0.0014, Log Rank
Statistical Analysis 3: Comparison: Placebo vs MDI 320 mcg/Day; Test type: Superiority or Other; p = 0.0062, Log Rank

7. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (TEAE)
Description: An adverse event was defined in the protocol as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an inability to carry out usual activities. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly/birth defect, or an important medical event that may not result in death, be life-threatening, or require hospitalization, but may jeopardize the patient and may require medical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Day 0 to Week 6
Population: The safety analysis set included all randomly assigned patients (ITT analysis set) who received at least 1 dose of study drug. In this analysis set, treatment was assigned based on the treatment patients actually received, regardless of the treatment to which they were randomly assigned.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BAI 320 mcg/Day | BAI 640 mcg/Day | MDI 320 mcg/Day
Number analyzed (Participants) | 107 | 108 | 105 | 105
Participants
  >=1 adverse event | 20 | 22 | 32 | 32
  >=1 mild TEAE | 10 | 10 | 18 | 20
  >=1 moderate TEAE | 9 | 11 | 10 | 11
  >=1 severe TEAE | 1 | 1 | 4 | 1
  >=1 treatment-related TEAE | 1 | 2 | 9 | 4
  >=1 serious TEAE | 0 | 0 | 2 | 0
  >=1 AE leading to withdrawal of study drug | 0 | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: Run-in Period: up to Day -30 to Day 0 Treatment Period: Day 0 to Week 6
Groups:
- Run-in Placebo: Pooled breath-actuated inhaler (BAI) and metered-dose inhaler (MDI) placebo groups. Participants were instructed to take 4 inhalations twice daily for up to 30 days of the single-blind Run-in Period.
- Placebo: Pooled breath-actuated inhaler (BAI) and metered-dose inhaler (MDI) placebo groups. Participants were instructed to take 4 inhalations twice daily for the 6 weeks of the double-blind Treatment Period.
- BAI 320 mcg/Day: Beclomethasone dipropionate breath-actuated inhaler (BAI), 4 inhalations (40 mcg/inhalation), twice daily for a total daily dose of 320 mcg for the 6 weeks of the double-blind Treatment Period.
- BAI 640 mcg/Day: Beclomethasone dipropionate breath-actuated inhaler (BAI), 4 inhalations (80 mcg/inhalation), twice daily for a total daily dose of 640 mcg for the 6 weeks of the double-blind Treatment Period.
- MDI 320 mcg/Day: Beclomethasone dipropionate metered-dose inhaler (MDI), 4 inhalations (40 mcg/inhalation), twice daily for a total daily dose of 320 mcg for the 6 weeks of the double-blind Treatment Period.
Arm/Group | Run-in Placebo | Placebo | BAI 320 mcg/Day | BAI 640 mcg/Day | MDI 320 mcg/Day
Serious Adverse Events (participants affected / at risk) | 1/713 | 0/107 | 0/108 | 2/105 | 0/105
Other Adverse Events (participants affected / at risk) | 0/713 | 3/107 | 5/108 | 5/105 | 10/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in Placebo (N=713) | Placebo (N=107) | BAI 320 mcg/Day (N=108) | BAI 640 mcg/Day (N=105) | MDI 320 mcg/Day (N=105)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in Placebo (N=713) | Placebo (N=107) | BAI 320 mcg/Day (N=108) | BAI 640 mcg/Day (N=105) | MDI 320 mcg/Day (N=105)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 5 (5) | 5 (5) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.